CLINICAL TRIAL: NCT03059901
Title: Caminamos: A Location-based Smartphone App for Latinas to Connect With Nearby Walking Partners
Brief Title: Caminamos: A Smartphone App to Connect With Walking Partners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klein Buendel, Inc. (Industry)
Collaborators: Stanford University (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R43MD009652 (NIH); R43MD009652-01 (NIH); 303 (Other: Klein Buendel, Inc.)
Record Dates: First submitted 2017-02-16; First posted 2017-02-23 (Actual); Results first posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-08

CONDITIONS: Physical Activity
Keywords: Physical Activity; Latina Women; Minority Health; Mobile Technology; Social Support
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- More App Notifications (Experimental): Participants receive more notifications than the Active Comparator group from the Caminamos app to walk.
  Interventions: Other: Caminamos App
- Normal App Notifications (Active Comparator): Participants receive less notifications than the Experimental group from the Caminamos app to walk.
  Interventions: Other: Caminamos App

INTERVENTIONS:
Other: Caminamos App — Mobile phone that encourages Latina women to walk together through social support.

SUMMARY:
Despite numerous interventions designed to increase physical activity, few are specifically tailored to Latinas, a population where higher rates of obesity, diabetes, and other chronic diseases are present. This proposed smartphone app will use location-based services to connect Latinas with one another in order to improve walking habits by increasing social support and decreasing perceived barriers, both of which are known to play a role in physical activity behaviors. In this Phase I research, surveys of potential end-users will determine interest in the app and focus groups will help shape a prototype of the app, which will be developed and tested to determine feasibility and functionality for a randomized Phase II intervention.

DETAILED DESCRIPTION:
Health disparities are high among Latinas. They are more likely to be overweight, diagnosed with diabetes, and physically inactive compared to their non-Hispanic White counterparts. Thus, interventions that target improving health access and ameliorating chronic diseases among Latinas are of high public health importance. Regular physical activity (PA) promotes physical and emotional well-being, yet PA interventions tailored for Latinas remain limited. Available data suggest that community-focused interventions produce improvements in physical activity (PA) and are well-received by Latinas especially when social and physical environments are considered (e.g., social support, safe walking areas, etc.). Research suggests that Latinos respond favorably to technological-based health interventions. Almost 90% of Latinos own a cellphone; 60% own a smartphone. Thus, health promotion interventions that can address Latinos' preferences regarding their physical and social environments while utilizing a preferred technology source (e.g., smartphone) could prove highly successful. One smartphone feature that offers great potential health promotion benefit is location-based services (LBS). LBS use geographic positioning to help users connect to their surrounding environment and to other users, thus providing them with real-time, user-specific information. This proposed project, ¡Caminamos!, will develop a smartphone app for use with 18-45 year old Latinas that uses LBS to connect women within geographically proximal neighborhoods as a way to provide social support for increased walking behaviors. Specific aims are: (1) gather input and evaluative feedback from an Expert Advisory Board (EAB) to help plan and assess the feasibility of creating the app; (2) build connections and gather input from Latino community leaders to assist in the conceptual development of the app through a Community Advisory Board (CAB); (3) conduct an online survey of a national sample of Latinas on their smartphone usage for health promotion, and interest in social networking and LBS technology features; (4) conduct iterative focus groups with Latinas age 18-45 years to guide development of app content, design, and aesthetics to fully develop a functioning prototype; and (5) conduct usability testing with Latinas to test the app's accuracy to establish users' location and connect users through the ¡Caminamos! system and users' use and satisfaction with the app. Few app-based health products are branded towards Latinas. ¡Caminamos! will address this unmet need in the marketplace. It will be the first smartphone app that uses location-based social networking to promote PA, and the only app of its kind targeted to Latinas. It will also expand upon what is known to be successful in Latino exercise engagement while simultaneously addressing key barriers to exercise. Phase I outcomes will provide the necessary framework and data for developing a full-scale app to be tested in a randomized clinical trial. In Phase III, we plan to market ¡Caminamos! directly to consumers in partnership with a company interested in expanding their brand outreach to a Latina population.

ELIGIBILITY:
Inclusion Criteria

* Eligibility criteria for online survey and focus groups is the ability to read and speak English or Spanish, female, consenting to inclusion in the study, self-identifying as Hispanic/Latina, and owning a smartphone.
* Eligibility criteria for usability testing is the ability to read and speak English or Spanish, female, consenting to inclusion in the study, self-identifying as Hispanic/Latina, owning a smartphone, and willing to use the app for a four-week period.

Exclusion Criteria:

* Exclusion criteria include being less than 18 years of age, being over 45 years of age, and being unable to speak or read English or Spanish.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Myers, PhD, Principal Investigator — Senior Scientist
Locations (2):
- United States (2):
  - Stanford University, School of Medicine, The Stanford Prevention Research Center, Palo Alto, California
  - Klein Buendel, Inc., Golden, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson M. Fact sheet: the state of Latinas in the United States. Center for American Progress. http://www.americanprogress.org/issues/race/report/2013/11/07/79167/fact-sheet-the-state-of-latinas-in-the-united-states/. December 7, 2013. Accessed: July 28, 2014.
- [Background] Adams PF, Kirzinger WK, Martinez ME. Summary health statistics for the u.s. Population: national health interview survey, 2011. Vital Health Stat 10. 2012 Dec;(255):1-110. PMID 25116371
- [Background] U.S.Department of Health & Human Services, Health Resources and Services Administration, Maternal and Child Health Bureau. Women's Health USA 2011. Rockville, Maryland: U.S. Department of Health and Human Services; 2011. http://www.mchb.hrsa.gov/whusa11/hstat/hshb/pages/201pa.html
- [Background] Warburton DE, Nicol CW, Bredin SS. Health benefits of physical activity: the evidence. CMAJ. 2006 Mar 14;174(6):801-9. doi: 10.1503/cmaj.051351. PMID 16534088
- [Background] Fisher KJ, Li F. A community-based walking trial to improve neighborhood quality of life in older adults: a multilevel analysis. Ann Behav Med. 2004 Dec;28(3):186-94. doi: 10.1207/s15324796abm2803_7. PMID 15576257
- [Background] Lee RE, Goldberg JH, Sallis JF, Hickmann SA, Castro CM, Chen AH. A prospective analysis of the relationship between walking and mood in sedentary ethnic minority women. Women Health. 2001;32(4):1-15. doi: 10.1300/J013v32n04_01. PMID 11548133
- [Background] Centers for Disease Control and Prevention. Physical activity and health. CDC Web site. http://www.cdc.gov/physicalactivity/everyone/health/. Accessed: July 28, 2014.
- [Background] Brown DW, Balluz LS, Heath GW, Moriarty DG, Ford ES, Giles WH, Mokdad AH. Associations between recommended levels of physical activity and health-related quality of life. Findings from the 2001 Behavioral Risk Factor Surveillance System (BRFSS) survey. Prev Med. 2003 Nov;37(5):520-8. doi: 10.1016/s0091-7435(03)00179-8. PMID 14572437
- [Background] Moadel AB, Shah C, Wylie-Rosett J, Harris MS, Patel SR, Hall CB, Sparano JA. Randomized controlled trial of yoga among a multiethnic sample of breast cancer patients: effects on quality of life. J Clin Oncol. 2007 Oct 1;25(28):4387-95. doi: 10.1200/JCO.2006.06.6027. Epub 2007 Sep 4. PMID 17785709
- [Background] Wilcox S, Bopp M, Oberrecht L, Kammermann SK, McElmurray CT. Psychosocial and perceived environmental correlates of physical activity in rural and older african american and white women. J Gerontol B Psychol Sci Soc Sci. 2003 Nov;58(6):P329-37. doi: 10.1093/geronb/58.6.p329. PMID 14614117
- [Background] Conn VS, Phillips LJ, Ruppar TM, Chase JA. Physical activity interventions with healthy minority adults: meta-analysis of behavior and health outcomes. J Health Care Poor Underserved. 2012 Feb;23(1):59-80. doi: 10.1353/hpu.2012.0032. PMID 22643462
- [Background] Juarbe T, Turok XP, Perez-Stable EJ. Perceived benefits and barriers to physical activity among older Latina women. West J Nurs Res. 2002 Dec;24(8):868-86. doi: 10.1177/019394502237699. PMID 12469724
- [Background] Ickes MJ, Sharma M. A systematic review of physical activity interventions in Hispanic adults. J Environ Public Health. 2012;2012:156435. doi: 10.1155/2012/156435. Epub 2012 Feb 8. PMID 22496702
- [Background] Lopez MH, Gonzalez-Barrera A, Patten E. Closing the digital divide : Latinos and technology adoption. Pew Research Center, Pew Hispanic Center. http://www.pewhispanic.org/files/2013/03/Latinos_Social_Media_and_Mobile_Tech_03-2013_final.pdf. March 7, 2013. Accessed: July 14, 2014.
- [Background] Zickuhr K. Three-quarters of smartphone owners use location-based services. Pew Internet & American Life Project. http://www.pewinternet.org/files/old-media/Files/Reports/2012/PIP_Location_based_services_2012_Report.pdf. May 11, 2012. Accessed: July 14, 2014.
- [Background] Albright CL, Pruitt L, Castro C, Gonzalez A, Woo S, King AC. Modifying physical activity in a multiethnic sample of low-income women: one-year results from the IMPACT (Increasing Motivation for Physical ACTivity) project. Ann Behav Med. 2005 Dec;30(3):191-200. doi: 10.1207/s15324796abm3003_3. PMID 16336070
- [Background] Smith A. Smartphone Ownership 2013 Update. Pew Research Internet Project. http://www.pewinternet.org/2013/06/05/smartphone-ownership-2013/. 2013. Accessed: July 14, 2014.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | More App Notifications | Normal App Notifications
Started | 30 | 30
Completed | 26 | 28
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | More App Notifications | Normal App Notifications | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.57 (7.86) | 33.0 (10.75) | 33.28 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 4 | 8
  More than one race | 21 | 18 | 39
  Unknown or Not Reported | 2 | 7 | 9
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: System Usability Questionnaire
Description: Participant perspective of program feasibility. Ten likert-type questions assessing user-friendliness of technology. Each question has five answer options that range from "Strongly Agree" to "Strongly Disagree". Scores range from 0-100. A score of 68 or above is considered above average. All scores averaged.
Time Frame: 4 weeks
Population: Although 60 women were enrolled, 6 women did not utilize the app during the trial. These 6 women (2 from More App Notifications and 4 from Normal App Notifications) were not included in the data analysis because they did not have data to analyze.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | More App Notifications | Normal App Notifications
Number analyzed (Participants) | 28 | 26
units on a scale | 60.54 (16.43) | 63.32 (16.67)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | More App Notifications | Normal App Notifications
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No